CLINICAL TRIAL: NCT02370849
Title: Cisplatin and S-1 With or Without Nimotuzumab for Patients With Previously Untreated Advanced Gastric Adenocarcinoma: a Single-center, Randomised, Open-label, Parallel-group, Controlled Phase 2 Clinical Trial
Brief Title: Cisplatin and S-1 With or Without Nimotuzumab in Untreated Advanced Gastric Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, yihebali chi, Assistant Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20150207
Record Dates: First submitted 2015-02-08; First posted 2015-02-25 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: Stomach Neoplasms
Keywords: nimotuzumab; gastric adenocarcinoma; Cisplatin; S-1; epidermal growth factor receptor
MeSH Terms: conditions — Stomach Neoplasms | interventions — nimotuzumab; Cisplatin; S 1 (combination)

ARMS (2):
- NCS (Experimental): nimotuzumab plus cisplatin and S-1
  Interventions: Drug: nimotuzumab; Drug: cisplatin; Drug: S-1
- CS (Active Comparator): cisplatin and S-1
  Interventions: Drug: cisplatin; Drug: S-1

INTERVENTIONS:
Drug: nimotuzumab — nimotuzumab 200mg infusion on day 1,8,15 every 3 weeks
  Arms: NCS
Drug: cisplatin — cisplatin: 30 mg/m2 iv. infusion on day 1, 2 every 3 weeks
Drug: S-1 — S-1: 40 mg/m2 bid , 2 weeks on, 1 week off ；

SUMMARY:
In this open-label, single-center, small sample size, randomised, parallel-group, controlled study, the investigators aim to assess efficacy and safety of addition of nimotuzumab to CS chemotherapy in patients with previously untreated advanced gastric adenocarcinoma. Sixty-two patients are required and randomly assigned (1:1) to each group.

The control regimen (CS chemotherapy) is recommended as the standard first-line regimen for advanced adenocarcinoma of the stomach or gastroesophageal junction in japan.

ELIGIBILITY:
Inclusion Criteria:

1. provision of written informed consent;
2. male or female; and aged ≥ 18 years;
3. Histologically verified, untreated, metastatic or locally advanced inoperable adenocarcinoma or signet ring cell carcinoma of the stomach or gastroesophageal junction;
4. At least one radiographically documented measurable lesion according to Response Evaluation Criteria In Solid Tumors Version 1.1(RECIST1.1) Criteria;
5. An Eastern Cooperative Oncology Group (ECOG) performance status of 0-2; and a life expectancy ≥ 3months;
6. No previous palliative chemotherapy;
7. Adequate function of vital organs: white blood cells (WBC) ≥ 4.0×109/L, neutrophils (ANA) ≥ 1.5 × 109/L, platelets ≥ 100 × 109/L, hemoglobin ≥ 90g/L (blood transfusion is permitted if necessary), serum bilirubin ≤ 1 times the upper normal limit (UNL), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 times the UNL, alkaline phosphatase (AKP) ≤ 5 times the UNL, creatinine (Cr) ≤ 1 times the UNL, normal electrocardiography (ECG).

Exclusion Criteria:

1. pregnant or lactating patients, or reproductive women without effective contraception;
2. Patients with only non-measurable disease: small lesions (longest diameter < 10mm or pathological lymph nodes with ≥ 10 to < 15mm short axis), Bone lesions, leptomeningeal disease, ascites, pleural or pericardial effusion, lymphangitic involvement of skin or lung; abdominal masses/abdominal organomegaly identified by physical exam that is not measurable by reproducible imaging techniques.
3. Symptomatic of brain metastasis;
4. Patients with clinically severe comorbidity including diabetes mellitus, hypertension, heart disease, or chronic active hepatitis (HBV carrier can be enrolled if circumstance permits );
5. No previous radiotherapy for measurable lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-10; Primary Completion 2012-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Objective response rate as measured by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) | 5 years

SECONDARY OUTCOMES:
Time to progression as measured by RECIST 1.1 | 5 years
Progression-free survival measured by RECIST 1.1 | 5 years
Treatment safety and toxicity as measured by Common Toxicity Criteria for Adverse Effects(CTCAE 3.0) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yihebali Chi, Doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China